CLINICAL TRIAL: NCT06471647
Title: Effects of Drugs on Stress Memories
Acronym: ETS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB23-1534
Record Dates: First submitted 2024-06-12; First posted 2024-06-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Delta-9-tetrahydrocannabinol (THC); Stress
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- placebo (Placebo Comparator): Dextrose capsules
  Interventions: Drug: Placebo
- 5 mg delta-9-tetrahydrocannabinol (THC) (Experimental): Marinol (dronabinol)
  Interventions: Drug: delta-9-tetrahydrocannabinol (THC) (5)
- 10 mg delta-9-tetrahydrocannabinol (THC) (Experimental): Marinol (dronabinol)
  Interventions: Drug: delta-9-tetrahydrocannabinol (THC) (10)

INTERVENTIONS:
Drug: delta-9-tetrahydrocannabinol (THC) (5) — 5 mg of THC
  Arms: 5 mg delta-9-tetrahydrocannabinol (THC)
Drug: Placebo — Placebo - dextrose
  Arms: placebo
Drug: delta-9-tetrahydrocannabinol (THC) (10) — 10 mg of THC
  Arms: 10 mg delta-9-tetrahydrocannabinol (THC)

SUMMARY:
There is evidence that cannabinoids, including delta-9-tetrahydrocannabinol (THC), reduce responses to acute stress and fear-related stimuli, but few studies have examined the effects of THC on memories of stressful experiences. The researchers hypothesize that THC will attenuate behavioral and physiological responses to negative valence stimuli, including memories of aversive experiences.

DETAILED DESCRIPTION:
The current study will use a between subject, randomized, placebo-controlled design to assess the effects of low doses of delta-9-tetrahydrocannabinol (THC) on stress memories. Healthy male and female participants (N=48) will be randomly assigned to one of the three drug conditions (5 mg THC [n=16], 10 mg THC [n=16], or placebo [n=16]). Each subject will participate in 3 sessions. In the first session, they will undergo the TSST procedure. Researchers will obtain ratings of subjective distress, heart rate variability, and cortisol levels to assess response to the stressor for each individual. On the second session, one week later, participants will receive either THC or placebo and they will then be presented with TSST-related cues during a stress-memory retrieval session.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 y/o
* BMI 19-29 kg/m2
* some prior experience with cannabis (used at least 4 times, no adverse experiences, and current use no more than once a week)

Exclusion Criteria:

* Current severe substance use disorder
* history of psychosis or mania
* Lack of English fluency
* Current DSM IV Axis I disorder
* Abnormal EKG
* Daily use of medications outside of contraception,
* Women who are pregnant or trying to become pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Change in emotional responses after stress memory cues compared to control cues after delta-9-tetrahydrocannabinol (THC) (5 mg, 10 mg) vs. placebo | baseline (5 minutes before memory task) and 20 seconds after each cue presentation during the task
  Using a visual analog scale participants will rate feelings of 'distress' 'arousal' and 'valence'. Scores range from 0-100 with higher scores indicating greater responses on particular items
Change in physiological responses after stress memory cue presentation compared to control cues | difference between values at baseline (5 minutes pre-task) and during 20 seconds of task cue presentations
  Researchers will assess changes in cardiac output (pre-ejection period) after presentation of cues. This will be measured in milliseconds. Lower values indicate greater sympathetic activation.

SECONDARY OUTCOMES:
Change in emotional responses one week later during non-drug retrieval session | 1 week after the first exposure they will complete the memory task again. The timeframe for assessing changes in emotional responses will be at baseline (5 minutes pre-memory task) and 20 seconds after each cue presentation
  Using a visual analog scale from 0-100 participants will rate feelings of 'distress' 'arousal' and 'valence' in a non-drug state. Scores range from 0-100 with higher scores indicating greater responses on particular items
Change in negative facial emotion expressions during cue presentation after THC (5 and 10 mg) vs placebo | During 20 seconds cue presentation
  Using facial expression model, researchers will assess changes in the intensity (0-1) of negative facial emotions during presentation of memory cues, comparing control vs. stress memory cues. higher values indicate greater intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States